CLINICAL TRIAL: NCT05294068
Title: Barriers to Physical Activity in Patients With Cognitive, Neuromotor or Sensory Impairments During Aging
Acronym: NO-BARRIERS
Status: Recruiting | Type: Observational
Sponsor: Institut de Sante Parasport Connecte Synergies (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-001
Record Dates: First submitted 2022-01-05; First posted 2022-03-24 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Disability or Chronic Disease Leading to Disablement
Keywords: Physical activities; Barriers; Disability
MeSH Terms: conditions — Motor Activity | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- All subjects with cognitive impairments
  Interventions: Other: standard of care for patients with cognitive impairments
- All subjects with neuromotor impairments
  Interventions: Other: standard of care for patients with neuromotor impairments
- All subjects with sensory impairments
  Interventions: Other: standard of care for patients with sensory impairments

INTERVENTIONS:
Other: standard of care for patients with cognitive impairments — clinical examination, radiological, biological and physiological examinations.
  Groups: All subjects with cognitive impairments
Other: standard of care for patients with neuromotor impairments — clinical examination, radiological, biological and physiological examinations.
  Groups: All subjects with neuromotor impairments
Other: standard of care for patients with sensory impairments — clinical examination, radiological, biological and physiological examinations.
  Groups: All subjects with sensory impairments

SUMMARY:
People with disabilities are less physically active than the general population. Their barriers to physical activity are multiple and include intrapersonal, organizational, societal and interpersonal reasons. Nevertheless, at present, the evolution of their barriers to physical activity and the short- and long-term impact of medical and medico-social treatments to limit them are unknown.

The aim of this study is to describe barriers to physical activity, or disability-related underperformance factors in competitive sports, in patients with cognitive, neuromotor or sensory impairments during aging.

DETAILED DESCRIPTION:
This is an ambispective, monocentric, cohort study of subjects with cognitive, neuromotor or sensory impairments followed in a Physical Medicine and Rehabilitation Department.

All consecutive eligible outpatient subjects consulting to the Parasport Health Unit of the Physical Medicine and Rehabilitation Department of our university hospital will be included. Clinical activities related to the Parasport Health Unit and performed outside the hospital will also be included.

Data will be collected from the patients' medical records, in particular data related to their clinical, radiological, biological and physiological examinations.

ELIGIBILITY:
Inclusion Criteria:

* Patients >= 6 years old ;
* Consulting to the Parasport Health Unit of the Physical Medicine and Rehabilitation Department of our university hospital ;
* Having a neuromotor, cognitive or sensory impairment ;
* No opposition to be enrolled in the study from the patient, or from a legally authorized close relative if the patient's state of health does not allow it, or from each of the holders of parental authority if a minor ;
* Affiliation to a social security scheme.

Exclusion Criteria:

* Under court protection.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with cognitive, neuromotor or sensory impairments.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2032-02-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Changes of barriers to physical activity during aging | through study completion, an average of 1 year
  Questionnaires assessing barriers and facilitators to physical activity (ex: BPAQ)

SECONDARY OUTCOMES:
Changes of physical activity level during aging | through study completion, an average of 1 year
  Questionnaires assessing physical activity levels (ex: PASPID)
Characteristics of medical and medico-social therapies implemented to limit barriers to physical activity | through study completion, an average of 1 year
  Number and description of medical and medico-social therapies
Characteristics of the medical and medico-social therapies implemented to limit disability-related underperformance factors for competitive sports | through study completion, an average of 1 year
  Number and description of medical and medico-social therapies
Characteristics of devices (orthoses, prostheses, etc.) and technical aids used to facilitate the practice of physical activity | through study completion, an average of 1 year
  Number and description of devices (orthoses and prostheses) and technical aids
Evolution of comorbidities during aging | through study completion, an average of 1 year
  Prevalence of comorbidities (e.g. obesity, diabetes, hypertension, sleep apnea, ...)
Evolution of exercise stress tests results during aging | through study completion, an average of 1 year
  Stress tests results

CONTACTS AND LOCATIONS:
Overall Officials: François Genêt, MD-PhD, Principal Investigator — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France; Vincent T Carpentier, MD-MSc, Study Director — Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, 92380 Garches, France
Locations (1):
- Department of Physical Medicine and Rehabilitation, Raymond Poincaré Hospital, AP-HP, Garches, France

IPD SHARING:
Plan to Share IPD: No